CLINICAL TRIAL: NCT00399919
Title: Safety and Efficacy pf Propionyl-L-Carnitine in Combination With Monitored Exercise Training in Peripheral Arterial Disease (Intermittent Claudication).
Brief Title: Safety and Efficacy of Propionyl-L-Carnitine in the Treatment of Peripheral Arterial Disease (Intermittent Claudication)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sigma-Tau Research, Inc. (Industry)
Collaborators: Colorado Prevention Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST 04-302
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2009-06

CONDITIONS: Peripheral Vascular Diseases; Intermittent Claudication
Keywords: Perhipheral Artery Disease; Claudication; Exercise; Intermittent Claudication due to Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Vascular Diseases; Intermittent Claudication; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLC (Experimental): Investigational drug
  Interventions: Drug: Propionyl-L-Carnitine; Drug: PLC
- Placebo (Placebo Comparator)
  Interventions: Drug: Propionyl-L-Carnitine; Drug: PLC

INTERVENTIONS:
Drug: Propionyl-L-Carnitine — 2 grams per day for six months
Drug: PLC — 2 grams/day for six months

SUMMARY:
Patients with peripheral artery disease have decreased blood flow to exercising muscle causing pain. This decreased blood flow to the muscle affects the level of acylcarnitines which in turn decreases the level of carnitine. Carnitine allows muscles to function properly. This study will test the safety and efficacy of Propionyl-L-Carnitine taken in combination with a monitored exercise training program.

DETAILED DESCRIPTION:
To test the hypothesis that Propionyl-L-Carnitine taken in combination with monitored exercise training may improve exercise performance the study will randomize male or female adults with peripheral artery disease and claudication to receive either Proprionyl-L-Carnitine or Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory outpatient who are able to exercise
* Intermittent claudication due to peripheral artery disease
* Willingness to participate in a monitored exercise training program

Exclusion Criteria:

* Pain at rest, ischemic ulcerations, gangrene of the lower extremity
* Peripheral Artery Disease of a non-atherosclerotic nature
* Any disease process other than PAD, that may interfere with performance during the treadmill test or prevent the subject from reaching their claudication-limited PWT
* Current participation in an exercise training program or previous participtation in a monitored exercise training program within 6 months of the screening visit.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2006-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Peak walking time | 6 months

SECONDARY OUTCOMES:
Claudication onset time, activity level and quality of life | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Carell, Principal Investigator — Western Suburban Cardiologists, Ltd.; Kenneth Morris, Principal Investigator — Durham VA Medical Center; Bruce Cutler, Principal Investigator — University of Massachusetts, Worcester; Robert McLafferty, Principal Investigator — SIU School of Medicine; Richard Powell, Principal Investigator — Dartmouth-Hitchcock Medical Center; Layne Yonehiro, Principal Investigator — Baptist Clinical Research; Karl Illig, Principal Investigator — University of Rochester; William Abernethy, Principal Investigator — Asheville Cardiology Associates; Michael Koren, Principal Investigator — Jacksonville Center For Clinical Research
Locations (9):
- United States (9):
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Baptist Clinical Research, Pensacola, Florida
  - Western Suburban Cardiologists, Ltd., LaGrange, Illinois
  - SIU School of Medicine, Springfield, Illinois
  - University of Massachusetts Medical Center, Worchester, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Rochester Medical Center, Rochester, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Durham VA Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Mays RJ, Wesselman CW, White R, Creager MA, Amato A, Greenwalt M, Hiatt WR. Automated Detection of Exercise Sessions in Patients With Peripheral Artery Disease: EVIDENCE FOR AN EXERCISE DOSE RESPONSE TO TRAINING. J Cardiopulm Rehabil Prev. 2021 May 1;41(3):176-181. doi: 10.1097/HCR.0000000000000553. PMID 33186199
- [Derived] Hiatt WR, Creager MA, Amato A, Brass EP. Effect of propionyl-L-carnitine on a background of monitored exercise in patients with claudication secondary to peripheral artery disease. J Cardiopulm Rehabil Prev. 2011 Mar-Apr;31(2):125-32. doi: 10.1097/HCR.0b013e3181f1fd65. PMID 20861750